CLINICAL TRIAL: NCT06159621
Title: Neoadjuvant/Phase 1 Study of CD40 Agonist (LVGN7409) and PD-1 Inhibitor (LVGN3616) in Patients With Resectable HPV-negative Mucosal Head/Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: CD40 Agonist and PD-1 Inhibitor in HNSCC
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 855063
Record Dates: First submitted 2023-11-16; First posted 2023-12-07 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Intervention Model Description: Patients will be assigned in an alternating fashion to Arm A (PD1 - LVGN 3616) or Arm B (PD1 LVGN 3616)+CD40 (LVGN 7409)). At a separate infusion visit after enrollment, patients in arm A or arm B will receive a single administration of LVGN3616 (300 mg.) or LVGN3616 (300 mg.) and LVGN7409 (1mg/kg), respectively. In case of patient drop-out after screening/consent and before drug administration, that slot will be assigned to the next available patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: PD1 (Active Comparator)
  Interventions: Drug: PD-1inhibitor - LVGN 3616
- Arm B: PD1 + CD40 (Active Comparator)
  Interventions: Drug: PD-1inhibitor - LVGN 3616; Drug: CD 40 Agonist - LVGN 7409

INTERVENTIONS:
Drug: PD-1inhibitor - LVGN 3616 — Administration of one dose of LVGN 3616 - 300mg. Commercially available PD-1 inhibitor may be substituted.
Drug: CD 40 Agonist - LVGN 7409 — Administration of one dose of LVGN 7409 - 1mg/kg
  Arms: Arm B: PD1 + CD40

SUMMARY:
Prospective, open-label, phase 1 study of CD40 agonist (LVGN7409) and PD-1 inhibition (LVGN3616 or nivolumab) in patients with resectable Human Papillomavirus (HPV)-negative mucosal head/neck squamous cell carcinoma (HNSCC). This protocol proposes to study the safety and immunological effects of LVGN7409, a CD40 agonistic antibody, when administered in combination with PD-1 inhibition prior to surgical resection.

DETAILED DESCRIPTION:
This will be a prospective, open-label, window of opportunity study of LVGN7409 and LVGN3616 (or nivolumab) in resectable HPV-negative HNSCC with co-primary endpoints of safety and T cell infiltration, and secondary endpoint of anti-tumor efficacy.

Doses of LVGN7409 and LVGN3616 (or nivolumab) are based on safety experience in prior and ongoing clinical trials. Dose escalation will not be conducted in this trial. The study is divided into the following treatment cohorts:

I. Arm A: PD1 [LVGN3616 (300mg) or nivolumab (240mg)] II. Arm B: PD1 [LVGN3616 (300mg) or nivolumab (240mg)] + CD40 [LVGN7409 (1mg/kg)]

Pre-Surgery and Surgery

1. Patients with potentially resectable HPV-negative HNSCC will be identified by H&N surgeons and study coordinator (clinic screening). Consent and enrollment will take place in H&N Surgery clinic by study investigators and/or the study coordinator.
2. Patients will need baseline non-Fine needle aspirate (FNA) tumor biopsy, either during standard of care exam under anesthesia (EUA) or via ultrasound-guided needle biopsy (prior archival non-FNA biopsy is acceptable as long as obtained within 6 months of screening).
3. Patients will be assigned in an alternating fashion to Arm A (PD1) or Arm B (PD1+CD40). At a separate infusion visit after enrollment, patients in arm A or arm B will receive a single administration of LVGN3616 (or nivolumab) or LVGN3616 (or nivolumab) and LVGN7409, respectively. In case of patient drop-out after screening/consent and before drug administration, that slot will be assigned to the next available patient.
4. Patients will be included in the primary endpoint calculations (safety) if they receive study drug. However, any patients unable to undergo planned surgery within 6 weeks will not contribute to the post-treatment immunologic sample analysis and this slot will be filled by a subsequent patient in order to achieve the goal of 10 paired samples in each arm. The maximum number of patients that can be replaced is 5.
5. After ~2 weeks (allowable range 6-42 days), patients will undergo planned surgical resection. Repeat imaging is not required.
6. Blood collection will occur on the day of drug administration prior to administration, 24-48 hours after administration, 1 week (+/-1 day) after administration, and on day of planned surgery. In person blood draws (D1, D7, etc.) can be waived in cases of transportation or logistical burden to the patient, at the discretion of the investigator.

Post-Surgery

1. Guideline-based standard of care post-surgical adjuvant therapies, as indicated based on pathological features on surgical resection, will occur as part of routine clinical care.
2. Post-operative visits will occur every 3 months (+/-4 weeks) after surgery up to 1 year, which will serve as End of trial (EOT) visit and final Adverse Event (AE) assessment. The following will be performed during each of these visits:

   1. Physical exam
   2. Laboratory monitoring
   3. AE assessment
   4. Concomitant medication review

ELIGIBILITY:
Inclusion Criteria:

* 1. Signed and dated written IRB-approved informed consent.
* 2. Age ≥18 years.
* 3. Body weight > 30kg
* 4. Human Papillomavirus (HPV)-negative histologically confirmed mucosal squamous cell head and neck cancer (oral cavity, oropharynx, larynx, hypopharynx) for which definitive surgery is planned. Sites other than oropharynx are assumed to be HPV negative unless specifically shown otherwise. Oropharynx HPV status can be determined through p16 or nucleic acid testing (ISH).
* 5. Tumor tissue sample (non-cytology specimen) available prior to Study Treatment, either via archived non-FNA (fine needle aspirate) tumor biopsy specimen or fresh biopsy
* 6. Life expectancy of at least 12 weeks.
* 7. Adequate bone marrow, hepatic, and renal function. ANC (Absolute Neutrophil Count) ≥ 1.5x109 cell/ml, platelets ≥75,000 /mm3, hemoglobin ≥9.0 g/dL, total serum bilirubin within 1.5 x upper limit of normal (ULN) unless Gilbert's, AST/ALT, within 2.5 x ULN, Albumin ≥3g/dL, and all tests performed within 4 weeks prior to administration of Study Treatment.
* 8. Eastern Cooperative Oncology Group (ECOG) with no clinically significant findings as assessed by the investigator.
* 9. ECOG performance status of 0-1.
* 10. Female patients of childbearing potential who are not abstinent and intend to be sexually active with a non-sterilized male partner must use at least 1 highly effective method of contraception from the time of screening throughout the total duration of the drug treatment and the drug washout period (90 days after therapy). Non-sterilized male partners of a female patient of childbearing potential must use male condom plus spermicide throughout this period. Female patients should also refrain from breastfeeding throughout this period.
* 11. Able and willing to comply with all study procedures.

Exclusion Criteria:

* 1. Prior history of Head and Neck Squamous Cell Carcinoma (HNSCC) for which patient has undergone surgery or radiation involving the current planned surgical site.

  2. Known history of hepatitis B or C with active viral replication. 3. Administration of any live vaccine within 28 days of first dose of study treatment.

  4. Prior anti-PD1 or CD40 agonist therapy. 5. Participation in another interventional clinical trial within 30 days before receiving first dose of study treatment. However, the subject may participate in observational studies.

  6. Any illness or condition that in the opinion of the investigator may affect the safety of the subject or the evaluation of any study endpoint.

  7. Current or prior use of immunosuppressive medication within 14 days before study treatment. The following are exceptions to this criterion:

  a. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection) b. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent.

  8. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of investigational product (IP).

  9. History of allogenic organ transplantation 10. Active or prior documented autoimmune disease. Examples include inflammatory bowel disease [e.g., colitis or Crohn's disease], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis], Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]. The following are exceptions to this criterion:
  1. Patients with vitiligo or alopecia
  2. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement or type 1 Diabetes Mellitus (DM) controlled with insulin.
  3. Any chronic skin condition that does not require systemic therapy.
  4. Patients without active autoimmune disease in the last 5 years may be included but only after consultation with the study physician.
  5. Patients with celiac disease controlled by diet alone. 11. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent 12. History of another active malignancy except for non-melanoma skin cancer, lentigo maligna or other carcinoma in situ 13. History of active primary immunodeficiency. Patients with Human Immunodeficiency Virus (HIV) with undetectable HIV viral loads by standard clinical assays are eligible.

     14. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2024-07-02 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
T cell frequency pre-treatment, as measured by immunohistochemistry (IHC) for CD8 on pre-treatment biopsy and resection tissue compared to T cell frequency post-treatment as measured by IHC for CD8 on biopsy and resection tissue post-treatment. | 1 year
Number of participants who undergo planned surgery within 6 weeks after drug administration | 6 weeks

SECONDARY OUTCOMES:
Pathological Response | 6 weeks
  Defined as the Percentage of the decrease in tumor resection bed replaced by necrotic tumor, histiocytes/giant cells fibrosis, and/or keratinous debris. Grading:
  * PTR0, <10% pathologic response
  * PTR1, 10%-49% pathologic response
  * PTR2, ≥50% pathologic response
Event free survival | 3 years
Progression free survival | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
No plan is in place